CLINICAL TRIAL: NCT07031193
Title: Instructional Influence: How Cueing Alters Foam Rolling Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Responsible Party: Principal Investigator, Kory Zimney, PT, DPT, PhD, Professor, University of South Dakota
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-25-143
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Foam Roller
Keywords: foam roller,; range of motion; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROM (Active Comparator): Foam rolling with instructions related to pain reduction
  Interventions: Procedure: Foam roller instructions for pain reduction; Procedure: Foam rolling for range of motion improvement
- Pain (Active Comparator): Foam rolling with Pain reduction instructions
  Interventions: Procedure: Foam roller instructions for pain reduction; Procedure: Foam rolling for range of motion improvement

INTERVENTIONS:
Procedure: Foam roller instructions for pain reduction — Foam rolling procedure with pain reduction instructions over hamstring muscle group
Procedure: Foam rolling for range of motion improvement — Foam rolling over hamstring muscle group with range of motion improvement instructions.

SUMMARY:
Foam rolling (FR) is a common tool and procedure used in rehabilitation. Previous research has demonstrated physical improvements in range of motion and subjective reductions in pain post-intervention. Most of the literature theorizes potential biophysical reasons for these changes, but definitive studies are lacking. Another potential mechanism for these improvements may be psychological.

The purpose of this study is to explore the psychological changes that occur in response to the instructions given to the patient and how these may influence the outcomes the individual receives while undergoing FR.

Different instructions will be given for the same technique of FR to see if there are differences in changes with pain and range of motion.

DETAILED DESCRIPTION:
Participants will receive one set of instructions that highlights the pain relieving properties of FR, while the other group will receive instructions on ability of FR to improve range of motion. Participants will be measured for range of motion and pain changes in both groups pre and post instruction and performing the identical technique of FR.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English and primary language

Exclusion Criteria:

* Current musculoskeletal injury of the lower limbs for which they are receiving medical care.
* Recent surgery to the lower limbs that has not been fully released for full participation by a medical provider.
* Use of any pain-relieving medications within the last 24 hours.
* Any medical condition that limits their perception of pain.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Straight leg raise Range of motion on dominate leg | from enrollment to the end of the session at 1 day
  Hamstring range of motion is measured with a standard goniometer on the dominant leg (the leg you would prefer to kick a ball with). Participant lying supine, the examiner assists with raising the leg straight (knee at 0 degrees extension) at the hip into flexion. Measure maximal hip flexion, with no change in knee extension, posterior pelvic tilt, or lumbar spine flexion. Goniometric measurements of hamstring length will then be measured with the stationary arm in line with the lateral midline of the pelvis, the axis of the goniometer will be placed on the greater trochanter of the hip, and the movement arm will be lined up with the midline of the lateral femur to the lateral epicondyle of the ipsilateral knee.
Pain pressure threshold of the hamstring muscle group | from enrollment to the end of the session at 1 day
  Use of a handheld algometer to assess pain pressure threshold. Application of pressure at the middle point of the hamstring on the dominant leg (the leg you would prefer to kick a ball with). The middle point is determined by the midway point measured from the ischial tuberosity and the knee joint line. Pressure is applied at a steady rate until the participant reports that the sensation of pressure changes from pressure to pain. Measurement in kg/cm2 will be recorded and the average of three measurements will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Dakota, Vermillion, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided